CLINICAL TRIAL: NCT04991948
Title: An Open-label, Phase Ib Study to Assess the Safety and Clinical Activity of CYAD-101 Administered Concurrently With FOLFOX Chemotherapy, Followed by Pembrolizumab Treatment, in Patients With Metastatic Colorectal Cancer
Brief Title: Study of Pembrolizumab Treatment After CYAD-101 With FOLFOX Preconditioning in Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-101-002; KEYNOTE-B79 (Other: Celyad Oncology)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — Folfox protocol; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYAD-101 with FOLFOX Infusion administered concurrently followed by pembrolizumab (Experimental)
  Interventions: Drug: CYAD-101; Drug: FOLFOX; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CYAD-101 — Allogeneic NKG2D-based CYAD-101 Chimeric antigen Receptor T-cells
Drug: FOLFOX — 5-FU, leucovorin and oxaliplatin
Drug: Pembrolizumab — Humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb)

SUMMARY:
The purpose of the CYAD-101-002 study is to assess the safety and clinical activity of CYAD-101 in patients with unresectable metastatic colorectal cancer administered concurrently with FOLFOX chemotherapy, followed by pembrolizumab treatment.

DETAILED DESCRIPTION:
This Study aims to provide insight into whether CYAD-101 administration concurrently with FOLFOX chemotherapy, followed by pembrolizumab treatment might be a treatment option for patients with unresectable metastatic colorectal cancer

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically proven metastatic adenocarcinoma of the colon or rectum.

   1. Confirmed metastatic unresectable adenocarcinoma of the colon or the rectum.
   2. Confirmed non-microsatellite instability high (non-MSI-H)/mismatch-repair proficient (pMMR) tumor status
   3. Unequivocal and measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
   4. Recurrent/progressing disease after at least one line of systemic therapy for metastatic disease which must include FOLFOX chemotherapy
   5. The patient is due to receive FOLFOX chemotherapy
   6. Neurotoxicity less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 from previous chemotherapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. Adequate organ, hepatic, renal, pulmonary and cardiac functions
4. Tumor biopsy at screening

Key Exclusion Criteria:

1. Any other investigational agent or device within 4 weeks of the first study treatment administration.
2. Any anticancer agent within 4 weeks of the first study treatment administration
3. Filgrastim (Granulocyte-Colony-Stimulating Factor [G-CSF]) or similar growth factors within 7 days of the first study treatment administration
4. Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
5. Prior radiotherapy within 2 weeks prior to the planned day for the first study treatment administration
6. Major surgery within 4 weeks before the planned day for the first study treatment administration
7. A live vaccine within 30 days prior to the planned day for the first study treatment administration
8. Uncontrolled intercurrent illness or serious uncontrolled medical disorder
9. Patients with history of (non-infectious) pneumonitis that require steroids or has current pneumonitis as assessed by chest imaging within 48 hours prior to first study treatment administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-08-21 (Estimated); Study Completion 2038-05-25 (Estimated)

PRIMARY OUTCOMES:
The Occurrence of Dose Limiting Toxicities (DLT) during the 'DLT reporting period' | Up to 73 days post first study treatment administration
  The occurrence of DLT during the 'DLT reporting period' is defined as the period from study enrollment on D1 (Visit 1) up to 3 weeks after first pembrolizumab treatment on D73 (Visit 14).
The objective response rate (ORR) at the tumor assessment on Day 94 [Visit 15]) | Up to 94 days post first study treatment administration
  The objective response rate (ORR) at the tumor assessment on Day 94 [Visit 15]), 6 weeks after the first pembrolizumab treatment administration.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Moffit Cancer Center, Tampa, Florida
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No